CLINICAL TRIAL: NCT04762407
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1903 in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1903
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROZE-103
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1 : Fasted state + HGP1910 + HGP1909, Period 2 : Fasted state + HCP1903
  Interventions: Drug: HGP1910; Drug: HGP1909; Drug: HCP1903
- Sequence 2 (Experimental): Period 1 :Fasted state + HCP1903, Period 2 : Fasted state + HGP1910 + HGP1909
  Interventions: Drug: HGP1910; Drug: HGP1909; Drug: HCP1903

INTERVENTIONS:
Drug: HGP1910 — Take it once per period.
Drug: HGP1909 — Take it once per period.
Drug: HCP1903 — Take it once per period.

SUMMARY:
An open-label, randomized, single-dose crossover study to evaluate the pharmacokinetics, safety and tolerability of HCP1903 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 29.9 kg/m^2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Cmax of Rosuvastatin | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
AUClast of Rosuvastatin | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
Cmax of Free Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
AUClast of Free Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation

SECONDARY OUTCOMES:
Cmax of Total Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
AUClast of Total Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
AUCinf of Rosuvastatin | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
Tmax of Rosuvastatin | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
t1/2 of Rosuvastatin | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
CL/F of Rosuvastatin | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
Vd/F of Rosuvastatin | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
AUCinf of Free Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
Tmax of Free Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
t1/2 of Free Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
CL/F of Free Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
Vd/F of Free Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
AUCinf of Total Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
Tmax of Total Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
t1/2 of Total Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
CL/F of Total Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation
Vd/F of Total Ezetimibe | pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No